CLINICAL TRIAL: NCT04619745
Title: Preventing Sedentary Lifestyles Among Children Born With Congenital Heart Defects; A Feasibility Study of Physical Activity After Surgical or Catheterization Intervention
Brief Title: A Feasibility Study of Physical Activity After Surgical or Catheterization Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Dr. Pat Longmuir, Senior Scientist, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20/67X
Record Dates: First submitted 2020-09-17; First posted 2020-11-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Congenital Heart Defect
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: In this model there is an intervention group and a wait-list control group. The intervention group will be receiving a 6-month, home-based, parent-led physical activity program, where as the control group will not receive this intervention until after the 12-month assessment.
Who Masked: Outcomes Assessor
Masking Description: A graduate student, blind to study group allocation, will conduct all assessments at each visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): All children enrolled in the study will complete five study visits. All participants will complete all outcome measures (including surveys, questionnaires, and motor skill assessments) at or after each 1-hour assessment visit. Children will be given an omni-directional accelerometer to wear on a waist-worn belt for 7 days after each visit to assess daily physical activity. The intervention group will complete individualized, parent-led, home and play-based activity plans for 6 months, beginning as soon as the child returns to the inpatient unit. The activities in the plan will be tailored to each phase of treatment (in hospital, discharge to week 7, week 8 to 6 months), follow a standardized format and provide content individualized to each child's age and previous visit assessments.
  Interventions: Other: Individualized Home and Play-Based Physical Activity Plans
- Wait List Control Group (Experimental): All children enrolled in the study will complete five study visits. After the first visit is complete, children will be randomized to either the intervention or wait-list control study group. Control participants will follow the same schedule of assessments at each visit, but the intervention will be provided between the 12-month and 16-month assessments. All participants will complete all outcome measures (including surveys, questionnaires, and motor skill assessments) at or after each 1-hour assessment visit. Children will be given an omni-directional accelerometer to wear on a waist-worn belt for 7 days after each visit to assess daily physical activity.
  Interventions: Other: Individualized Home and Play-Based Physical Activity Plans

INTERVENTIONS:
Other: Individualized Home and Play-Based Physical Activity Plans — Play-based, parent led interventions optimized to support age appropriate physical activity, and motor skills among young children with congenital heart defects.

SUMMARY:
This feasibility study will assess whether a 6-month, home-based, parent-led physical activity program, completed after surgical or catheterization treatment, enables young children with congenital heart defects (CHD) to achieve the recommended 180 minutes of daily physical activity. This study includes comprehensive measures of motor skill and physical activity, intervening at a very young age, and targeting the high risk status for sedentary lifestyles of children with CHD. This study will provide essential data on patient recruitment, data collection procedures, the proposed physical activity intervention and resources required to enable the design of a randomized controlled trial (RCT) to evaluate play-based, parent-delivered interventions optimized to support age-appropriate physical activity and motor skills among young children with CHD.

DETAILED DESCRIPTION:
This study addresses the issue that congenital heart defect (CHD) treatment in infants and young children causes limitations that reduce active play opportunities, delaying motor skill development, and preventing active lifestyle habits from being established in early childhood. Recent research has shown that the most sedentary children assessed in infancy continue to be the most sedentary children at school age. This suggests that an effective intervention to enhance active play and prevent sedentary lifestyles must target children with CHD in infancy.

The investigators hypothesize that intervening during the treatment (via surgery or catheterization) and post-treatment recovery phase would be optimal for changing physical activity habits among young children with CHD. Thus, this feasibility study will assess whether a 6-month, home-based, parent-led physical activity program, completed after surgical or catheterization treatment, enables young children with CHD to achieve the recommended 180 minutes of daily physical activity.

This study includes comprehensive measures of motor skill and physical activity, intervening at a very young age, and targeting the high risk status for sedentary lifestyles of children with CHD. This study will provide essential data on patient recruitment, data collection procedures, the proposed physical activity intervention and resources required to enable the design of an RCT to evaluate play-based, parent-delivered interventions optimized to support age-appropriate physical activity and motor skills among young children with CHD. Children who are scheduled for cardiac surgery or catheterization will be recruited during the study recruitment period. The estimated initial sample size of recruited patients is 56, however factoring in withdrawal rate, it is expected that feasibility data will be obtained for 48 participants. Eligible participants who agree to be contacted by a member of the research team will have the study explained to them in full detail and will sign a consent form if desired. All children in this study will complete five study visits. The first study visit will consist of gaining the patient's consent and performing a baseline assessment on the patient. After the first visit is complete, children will be randomized to either the intervention or wait-list control study group. Control participants will follow the same schedule of assessments but they will be on a "wait list" for the intervention, which will be provided after the 12-month assessment has been completed.The first visit will occur during the mandatory pre-treatment clinic visit, which is typically 1-2 weeks prior to treatment. Visits #2, #3, #4 and #5 will occur 7 weeks and 6, 12 and 16 months after treatment. All participants will complete all outcome measures and assessments at or after each visit. Children will be given an omni-directional accelerometer to wear on a waist-worn belt for 7 days after each visit, to assess daily physical activity. Movement skills will be assessed with the Peabody Motor Development Scales (version 2). Parents will complete a demographic questionnaire, the Pediatric Quality of Life Inventory (PedsQL51) proxy report for toddlers/young children, the Social Skills Checklist, Parenting Stress Index, and parents of children 4 years or younger will complete the Infant Quality of Life assessment. The child's medical history will be extracted from the medical record.

Each child receiving CHD treatment randomized to the intervention group will be provided with 6 months of parent-led, home and play-based activity plans. The activities in the plan will be tailored to each phase of treatment (in hospital, discharge to week 7, week 8 to 6 months), follow a standardized format and provide content individualized to each child's age and previous visit assessments. The in-hospital intervention will begin when the child returns to the regular hospital ward from the ICU. Play activities will focus on maintaining or regaining range of motion and supporting midline crossing. Resumption of the motor skills and mobility demonstrated prior to treatment will be encouraged once all treatment equipment has been removed. From time of discharge to the week 7 follow up, a range of motion and mobility intervention will be provided. It will be similar to the in-hospital plan but with the addition of lower body mobility activities to encourage movement skill development. Upper body weight bearing and lifting activities are restricted for children undergoing surgical treatment until the week 7 evaluation. The research assistant will monitor/adjust the child's physical activity on a weekly basis until activity is unrestricted. Once physical activity is unrestricted, parent-led, home and play-based weekly plans will be designed by the research assistant to encourage active lifestyle habits during the time between the week 7 and 6 month visit. Each plan will be individualized to the child's age and assessment results. A new set of progressive activity plans will be provided every four weeks until the end of the intervention (6 month visit), using parent feedback regarding the child's progress and the attainment of age-appropriate motor skills. The research assistant will also educate parents about their child's assessed and desired level of daily physical activity and support parents as they implement the activity plans at home. The research assistant on the project will see children daily during their hospitalization, working with parents to implement the child's personal activity plan. Collaborative implementation will enable the research assistant to ensure accurate performance of target movements and answer parent questions. The research assistant will track all data, study details and patient interactions.

ELIGIBILITY:
Inclusion Criteria

1. Female or male at least 3 months of age but not more than 72 months of age (upper age limit for valid Peabody Motor Development Scales-2 assessment)
2. Receiving elective treatment via cardiac surgery or catheterization intervention for CHD at the Children's Hospital of Eastern Ontario.

Exclusion Criteria

1. Genetic conditions or physical disabilities impacting motor development (e.g., Down syndrome)
2. Emergency treatment for child in critical condition
3. Medical care not compatible with study assessments
4. No independent limb movement.

Ages: 3 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of patient recruitment measured as # surgical patients, # cath patients, # eligible, # approached, # willing to enroll, # withdrawn | 18 months
  Monthly: # surgical patients, # cath patients, # eligible, # approached, # willing to enroll, # withdrawn
Feasibility of patient randomization measured as # of patients/parents willing to randomize | 18 months
  Monthly: # of patients/parents willing to randomize
Feasibility of data collection procedures measured as % of patients with complete pretreatment data | 18 months
  % of patients with complete pretreatment data; days available prior to treatment for baseline data collection; % of parents able to complete child accelerometer wear for 7 days; % of control and intervention who complete all data sessions; frequency of missing data

SECONDARY OUTCOMES:
Retention and follow up rates measured as # participants retained in study; # follow up sessions complete | 18 months
  End of Study: # participants retained in study; # follow up sessions complete
% compliant with intervention and rate of adherence | 18 months
  Per follow up call: % of participants that completed each intervention, % of sessions completed weekly

OTHER OUTCOMES:
Clarity of inclusion/exclusion criteria measured as # requiring MD consult for eligibility | 18 months
  Monthly: # inclusion/exclusion is clear, # requiring MD consult for eligibility, # ineligible after baseline, # of patients excluded who could participate
healthcare professionals facilitate recruitment measured as # of days for MD approval | 18 months
  Monthly: # of days prior to treatment schedule is set, time to screen eligibility, # of days for MD approval, # of days for circle of care contact, # of days for family contact/consent
study time and burden measured as parent rating of time and burden (100mm visual analogue scale) | 18 months
  Per visit: Parent rate a) time and b) burden (100mm visual analogue scale) End of study: Ratings of time and burden by healthcare professionals
intervention time and burden measured as parent rating of time and burden (100mm visual analogue scale) | 18 months
  Per visit: Parent rate time and burden (1 to 100 scale, higher number meaning more burden) and provide qualitative feedback End of study: Ratings of time and burden and qualitative feedback from healthcare professionals
Resources to conduct the RCT measured as staff time required | 18 months
  staff time required to identify, consent and follow patients; space available for baseline testing; kinesiologist time to create and support interventions

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ginsburg KR; American Academy of Pediatrics Committee on Communications; American Academy of Pediatrics Committee on Psychosocial Aspects of Child and Family Health. The importance of play in promoting healthy child development and maintaining strong parent-child bonds. Pediatrics. 2007 Jan;119(1):182-91. doi: 10.1542/peds.2006-2697. PMID 17200287
- [Background] Bar-Or O, Rowland TW. Habitual activity and energy expenditure in the healthy child. Pediatric Exercise Medicine: From Physiologic Principles to Health Care Application. Champaign, IL: Human Kinetics; 2004. p. 64-7.
- [Background] Klavora P. Foundations of Exercise Science. Toronto, Ontario: Sport Books Publisher; 2004.
- [Background] Centers for Disease Control. Physical activity for everyone: The importance of physical activity. 2005; Available at: URL: http://www.cdc.gov/nccdphp/dnpa/physical/importance/index.htm. Accessed August 9, 2007.
- [Background] Timmons BW, Naylor PJ, Pfeiffer KA. Physical activity for preschool children--how much and how? Can J Public Health. 2007;98 Suppl 2:S122-34. PMID 18213943
- [Background] Longmuir PE, McCrindle BW. Physical activity restrictions for children after the Fontan operation: disagreement between parent, cardiologist, and medical record reports. Am Heart J. 2009 May;157(5):853-9. doi: 10.1016/j.ahj.2009.02.014. PMID 19376311
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Project DATA. Social Skills Checklist. 2007. St. Louis, University of Washington. 7-20-2019. Ref Type: Serial (Book,Monograph)
- [Background] Abidin RR. Parenting Stress Index. 3rd ed. Odessa, Florida: Psychological Assessment Resources, Inc.; 1990.
- [Background] Stieber NA, Gilmour S, Morra A, Rainbow J, Robitaille S, Van Arsdell G, McCrindle BW, Gibson BE, Longmuir PE. Feasibility of improving the motor development of toddlers with congenital heart defects using a home-based intervention. Pediatr Cardiol. 2012 Apr;33(4):521-32. doi: 10.1007/s00246-011-0144-0. Epub 2011 Nov 25. PMID 22116604
- [Derived] Ramanan N, Lee S, Maharajh G, Webster R, Longmuir PE. Preventing sedentary lifestyles among young children born with congenital heart defects: A feasibility study of physical activity rehabilitation after surgical or catheterization intervention. PLoS One. 2023 Aug 18;18(8):e0284946. doi: 10.1371/journal.pone.0284946. eCollection 2023. PMID 37594946